CLINICAL TRIAL: NCT05663047
Title: Prevent It 2.0/GPP - Internet Mediated Cognitive Behavioral Therapy to Reduce the Risk of Committing Child Sexual Abuse - Global Perpetrator Prevention Project
Brief Title: Prevent It 2.0/GPP -iCBT to Reduce the Risk of Committing Child Sexual Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Royal Ottawa Mental Health Centre (Other); Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Principal Investigator, Christoffer Rahm, MD, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Prevent It 2.0/GPP
Record Dates: First submitted 2022-11-28; First posted 2022-12-23 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-10

CONDITIONS: Pedophilia
Keywords: Child sexual abuse; Pedophilic disorder; Preventive psychiatry; Internet based intervention; Cognitive behavioral therapy; Waitlist
MeSH Terms: conditions — Pedophilia | interventions — Waiting Lists

STUDY DESIGN:
Intervention Model Description: An academically initiated randomized controlled clinical trial where Prevent It 2.0 is compared with waitlist control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prevent It 2.0 (Experimental)
  Interventions: Other: Prevent It 2.0
- Waitlist (Active Comparator)
  Interventions: Other: Waitlist

INTERVENTIONS:
Other: Prevent It 2.0 — A free, anonymous, internet-delivered, therapist assisted, cognitive behavioral therapy (CBT) intervention
  Arms: Prevent It 2.0
Other: Waitlist — Participants in the waitlist control will wait thirteen weeks before starting active treatment. While on the waitlist, participants will respond to questions about ongoing problematic sexual behavior.
  Arms: Waitlist

SUMMARY:
Child sexual abuse is a large-scale global problem, and with the internet and communication technologies enabling new ways to sexually abuse children, the problem is drastically increasing.

Prevent It is a free, anonymous, internet-delivered, therapist assisted, cognitive behavioral therapy (CBT) intervention for individuals concerned about their sexual urges or behaviors involving children. The treatment program is based on many years of clinical experience from working with this patient group, results from several previous research projects.

Using the scientifically rigorous design of a randomized controlled trial with waitlist control, we want to evaluate Prevent It 2.0 - an updated cognitive behavioral therapy treatment for individuals who are concerned about their sexual urges regarding children.

The study design is an academically initiated randomized controlled clinical trial where Prevent It 2.0 is compared with waitlist control. Participants in the waitlist control will wait thirteen weeks before starting active treatment. While on the waitlist, participants will respond to questions about ongoing problematic sexual behavior.

Recruitment will be carried out through multiple channels, and takes place on both "Darknet" and "Clearnet". All contact with participants, the treatment, evaluations, and termination of the contact, is conducted via the online treatment platform Iterapi, designed specifically for clinical trials of Internet-mediated CBT.

The treatment contains nine modules over thirteen weeks and the content of the therapy is classic CBT.

ELIGIBILITY:
Inclusion Criteria:

* concern about sexual urges regarding children
* Informed consent to participate

Exclusion Criteria:

* Participants with a severe psychiatric illness (such as high acute suicide risk or severe substance abuse)
* Participants that are judged to have a limited understanding of the languages that the treatment is delivered in (English)
* Lack serious intention to participate (assessed by the researcher/therapist during the intake interview, which lasts approximately one hour)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2022-11-25 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2025-02-11 (Actual)

PRIMARY OUTCOMES:
1. Is Prevent It 2.0 effective in reducing participants' urges to act on sexual behaviors involving children, as measured by the SSAS (Sexual Symptom Assessment Scale)?involving children | Up to 13 weeks
  Sexual Symptom Assessment Scale, The range is 0 to 48, with 0 indicating no symptoms and 48 indicating severe symptoms.

SECONDARY OUTCOMES:
Is Prevent It 2.0 effective in reducing participants' sexual behaviors involving children, as measured by the Sexual Child Molestation Risk Assessment (the SChiMRA+) Part B? | Up to 13 weeks
  The Sexual Child Molestation Risk Assessment, there's no scoring system at the moment. It's all item-by-item. But for all items, higher values are worse (e.g., more hours watching CSAM, more motivation to interact with children, etc).

OTHER OUTCOMES:
Is Prevent It 2 safe from a negative side effects perspective, as measured by the Negative Effects Questionnaire (NEQ-20)? | Up to 13 weeks
  NEQ-20 taps the occurrence (binary, yes or no) and severity (on a 5-point Likert scale 0-4, ranging from not at all to extremely) of 20 statements regarding negative effects of psychological treatment and ends with one free-text question. For each statement answered with yes , the respondent also reports whether they believe the negative effect is caused by "the treatment I received" or "other circumstances". Maximum score = 80, Minimum score = 0.
Comparisons of attrition rates in active arm and waitlist in Prevent It 2, to active arm and placebo in Prevent It 1? | Up to 13 weeks
Comparisons of SChiMRA in active arm and waitlist in Prevent It 2, to active arm and placebo in Prevent It 1? | Up to 13 weeks
Comparisons of NEQ-20 in active arm and waitlist in Prevent It 2, to active arm and placebo in Prevent It 1? | Up to 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christoffer Rahm, MD, Principal Investigator — Karolinska Institutet
Locations (1):
- CPF - centrum för psykiatriforskning., Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in each respective article, after deidentification (text, tables, figures and appendices). Fully deidentified participant data will be shared in a public repository without demographic information. Data with demographic information will be shared with an approved data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: For data shared through a data access agreement, beginning 3 months and ending 5 years following each article publication. Data shared in a public repository will be available immediately following each article publication and will be available for at least 5 years.
Access Criteria: For data that contain demographic information, investigators who provide a methodologically sound proposal, and whose proposed use of the data has been approved by an independent review committee identified for this purpose. Any researcher may access the version of the data available in a public repository.
  * For what types of analyses? To achieve aims in the approved proposal and for meta-analysis
  * By what mechanism will data be made available? Proposals should be directed to Christoffer.rahm@ki.se. To gain access to the data with demographic information, data requesters will need to sign a data access agreement. Data will be made available digitally via a secure data transfer facility provided by Karolinska Institute. Fully deidentified data without demographics will be made available on the Open Science Framework (osf.io).
URL: https://osf.io/y2dc4/?view_only=